CLINICAL TRIAL: NCT06496542
Title: Renal Oxygen Consumption, Insulin Sensitivity, and Daily Caloric Restriction in Autosomal Dominant Polycystic Kidney Disease (EXPLORE Study)
Brief Title: Renal Oxygen Consumption, Insulin Sensitivity, and Daily Caloric Restriction in ADPKD
Acronym: EXPLORE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Nutrition Obesity Research Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-0979; P30DK048520 (NIH)
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Autosomal Dominant Polycystic Kidney
Keywords: Kidney Disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Kidney Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Caloric Restriction (Experimental): The daily caloric restriction group will participate in a 2-year, group-based, behavioral weight loss intervention based on a 30% reduction in caloric intake and increased physical activity.
  Interventions: Behavioral: Daily caloric restriction
- Other: Standard Advice Control (Other): The standard advice control group will receive an initial consultation with a registered dietician regarding current clinical recommendations for ADPKD without subsequent counseling sessions.
  Interventions: Other: Standard advice control

INTERVENTIONS:
Behavioral: Daily caloric restriction — Weight loss based on daily caloric restriction and increased physical activity
  Arms: Daily Caloric Restriction
Other: Standard advice control — Initial nutrition consultation without subsequent counseling
  Arms: Other: Standard Advice Control

SUMMARY:
The proposed research is a pilot study assessing kidney oxidative metabolism and insulin sensitivity after a 2-year weight loss intervention in those with autosomal dominant polycystic kidney disease who are overweight or obese.

DETAILED DESCRIPTION:
Autosomal dominant polycystic kidney disease (ADPKD) is the most commonly inherited progressive kidney disease. Overweight and obese phenotypes have been associated with disease progression in early-stage ADPKD. Daily caloric restriction (DCR, 34% restriction per day from baseline weight maintenance requirements) may aid in weight loss and ultimately slow ADPKD disease progression. Weight loss via DCR may cause alterations in kidney oxidative metabolism and insulin sensitivity that can affect ADPKD disease progression. This study aims to assess kidney oxidative metabolism via 11C-acetate PET scan protocol and insulin sensitivity via hyperinsulinemic-euglycemic clamp by leveraging an ongoing R01-funded trial (NCT04907799) in DCR (n=10) vs. control (n=10) groups at baseline (BSL) and 2 years. The study will utilize the clinical outcome measures performed in the parent trial to address the subsequent novel aims: Aim 1: Compare kidney oxidative metabolism and insulin sensitivity at BSL and 2 years in adults with ADPKD. Aim 2: Define the relations among changes in kidney oxidative metabolism, insulin sensitivity, total kidney volume, and weight over 2 years. Currently, it is unknown if weight loss via DCR modifies renal energy expenditure and substrate utilization.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* ADPKD diagnosis based on the modified Pei-Ravine criteria
* Body-mass index of 25-45 kg/m^2
* Estimated glomerular filtration rate ≥ 30 mL/min/1.73m^2
* Total kidney volume (htTKV) > 600 mL, calculated from a previous kidney ultrasound or magnetic resonance imaging performed within the last 12 months
* Access to the internet with video chat capabilities
* No plans for extended travel (>2 weeks) without internet access during the 12-month intensive period
* Not currently participating in or planning to participate in any formal weight loss or physical activity program, or another interventional study
* Ability to provide informed consent

Exclusion Criteria:

* Diabetes mellitus
* Current smokers or history of smoking in the past 12 months
* Alcohol dependence or abuse
* History of hospitalization or major surgery within the last 3 months
* Untreated dyslipidemia
* Uncontrolled hypertension
* Pregnancy, lactation, or unwillingness to use adequate birth control
* Cardiovascular disease, peripheral vascular disease, or symptoms suggestive of cardiovascular disease: chest pain, shortness of breath at rest or with mild exertion, syncope
* Abnormal resting electrocardiogram (ECG): serious arrhythmias, including multifocal premature ventricular contractions (PVC's), frequent PVC's (defined as 10 or more per min), ventricular tachycardia (defined as runs of 3 or more successive PVC's), or sustained atrial tachyarrhythmia; 2nd or 3rd degree A-V block, QTc interval > 480 msec or other significant conduction defects
* Significant pulmonary disease including: chronic obstructive pulmonary disease, interstitial lung disease, cystic fibrosis, or uncontrolled asthma
* Regular use of prescription or over-the-counter medications that may affect weight, appetite, food intake, or energy metabolism
* History of clinically diagnosed eating disorder including: anorexia nervosa, bulimia, binge eating disorder
* Weight loss of >5% in the past 3 months for any reason except post-partum weight loss; weight gain >5% requires assessment by PI
* Major psychiatric disorder (e.g., psychosis, schizophrenia, mania, bipolar disorder) or current severe depression, based on DSM-IV-TR criteria for Major Depressive Episode, which in the opinion of the Study MD would interfere with ability to adhere to dietary interventions)
* Inability to cooperate with or clinical contraindication for magnetic resonance imaging, including: severe claustrophobia, implants, devices, or non-removable body piercings
* Previous obesity treatment with surgery or weight loss device, except: (1) liposuction and/or abdominoplasty if performed > 1 year before screening, (2) lap banding if the band has been removed > 1 year before screening, (3) intragastric balloon if the balloon has been removed > 1 year before screening (4) duodenal-jejunal bypass sleeve, if the sleeve has been removed > 1 year before screening or 5) AspireAssist or other endoscopically placed weight loss device if the device has been removed > 1 year before screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in renal oxygen consumption | Baseline, 24-months
  Renal oxygen consumption will be assessed by a PET/CT scan using 11-C acetate
Change in insulin sensitivity | Baseline, 24-months
  Insulin sensitivity will be assessed by a hyperinsulinemic-euglycemic clamp

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado- Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039